CLINICAL TRIAL: NCT03070886
Title: Phase II-III Trial of Adjuvant Radiotherapy and Androgen Deprivation Following Radical Prostatectomy With or Without Adjuvant Docetaxel
Brief Title: Antiandrogen Therapy and Radiation Therapy With or Without Docetaxel in Treating Patients With Prostate Cancer That Has Been Removed by Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU002; NCI-2016-00963 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU002; NRG-GU002 (Other: NRG Oncology); NRG-GU002 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2016-12-30; First posted 2017-03-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Stage I Prostate Adenocarcinoma AJCC v7; Stage II Prostate Adenocarcinoma AJCC v7; Stage III Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — bicalutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Docetaxel; Congresses as Topic; Radiation; Flutamide; Salicylic Acid; Goserelin; Leuprolide; luprolide acetate gel depot; nilutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (androgen deprivation therapy, EBRT) (Active Comparator): Patients receive androgen deprivation therapy comprising leuprolide acetate, goserelin acetate, degarelix, bicalutamide, flutamide, or nilutamide for 6 months. Beginning 8 weeks after the start of androgen deprivation therapy, patients receive EBRT for 7.5 weeks.
  Interventions: Drug: Bicalutamide; Drug: Degarelix; Radiation: External Beam Radiation Therapy; Drug: Flutamide; Drug: Goserelin; Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Drug: Leuprolide; Drug: Leuprolide Acetate; Drug: Nilutamide
- Arm II (androgen deprivation therapy, EBRT, docetaxel) (Experimental): Patients receive androgen deprivation therapy and EBRT as in Arm I. Within 4-6 weeks after completion of radiation therapy, patients receive docetaxel IV over 1 hour on day 1 of every 21 days for 6 cycless in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Bicalutamide; Drug: Degarelix; Drug: Docetaxel; Radiation: External Beam Radiation Therapy; Drug: Flutamide; Drug: Goserelin; Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Drug: Leuprolide; Drug: Leuprolide Acetate; Drug: Nilutamide

INTERVENTIONS:
Drug: Bicalutamide — Given orally (PO)
  Other Names: Casodex; Cassotide; Cosudex; ICI 176,334; ICI 176334; Utamide
Drug: Degarelix — Given IM
  Other Names: ASP 3550; ASP-3550; ASP3550; FE 200486; FE-200486; FE200486; Firmagon
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm II (androgen deprivation therapy, EBRT, docetaxel)
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Drug: Flutamide — Given PO
  Other Names: 4'-Nitro-3'-trifluoromethylisobutyranilide; Apimid; Cebatrol; Chimax; Cytomid; Drogenil; Euflex; Eulexine; Flucinom; Flucinome; Flugerel; Fluken; Flulem; FLUT; Fluta-Gry; Flutabene; Flutacan; Flutamex; Flutamin; Flutan; Flutaplex; Fugerel; Grisetin; Niftolide; Oncosal; Profamid; Propanamide, 2-Methyl-N-(4-nitro-3-(trifluoromethyl)phenyl)-; Prostacur; Prostadirex; Prostica; Prostogenat; Sch 13521; Tafenil; Tecnoflut; Testotard
Drug: Goserelin — Given IM
  Other Names: ICI-118630
Drug: Goserelin Acetate — Given IM
  Other Names: ZDX; Zoladex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leuprolide — Given intramuscularly (IM)
  Other Names: Leuprorelin
Drug: Leuprolide Acetate — Given IM
  Other Names: A 43818; A-43818; A43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Fensolvi; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Luprodex Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Lutrate; Procren; Procrin; Prostap; TAP 144; TAP-144; TAP144; Trenantone; Uno-Enantone; Viadur
Drug: Nilutamide — Drug
  Other Names: Anandron; Nilandron; RU-23908

SUMMARY:
This randomized phase II/III trial studies docetaxel, antiandrogen therapy, and radiation therapy to see how well it works compared with antiandrogen therapy and radiation therapy alone in treating patients with prostate cancer that has been removed by surgery. Androgen can cause the growth of prostate cells. Antihormone therapy may lessen the amount of androgen made by the body. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving antiandrogen therapy and radiation therapy with or without docetaxel after surgery may kill any remaining tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the benefit of docetaxel as measured by improvement in freedom from progression (phase II) and subsequently metastasis free survival (phase III) when given in combination with radiation and androgen deprivation in treatment of high risk prostate cancer post-radical prostatectomy.

SECONDARY OBJECTIVES:

I. To assess overall survival. II. To assess local time to progression. III. To assess undetectable prostate-specific antigen (PSA) with a non-castrate testosterone at 2.5 years post treatment.

IV. To assess the utility of genomic profiling in making adjuvant therapy decisions post-prostatectomy.

V. To assess toxicity of docetaxel in the post-operative setting when combined with radiation and androgen deprivation therapy.

VI. To assess treatment response by genomically defined sub-groups of prostate cancer patients.

EXPLORATORY OBJECTIVE:

I. To optimize quality assurance methodologies and processes for radiotherapy and imaging, with machine learning strategies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive androgen deprivation therapy comprising leuprolide acetate, goserelin acetate, degarelix, bicalutamide, flutamide, or nilutamide for 6 months. Beginning 8 weeks after the start of androgen deprivation therapy, patients receive external beam radiation therapy (EBRT) for 7.5 weeks.

ARM II: Patients receive androgen deprivation therapy and EBRT as in Arm I. Within 4-6 weeks after completion of radiation therapy, patients receive docetaxel intravenously (IV) over 1 hour on day 1 of every 21 days for 6 cycles in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for 3 years, and then yearly.

ELIGIBILITY:
Inclusion Criteria:

* Patients post-prostatectomy with baseline Gleason >= 7 (per prostatectomy pathology)
* Baseline PSA prior to start of androgen deprivation therapy nadir >= 0.2 ng/ml (post-operative value is never undetectable) obtained prior to step 1 registration
* Baseline testosterone level obtained post-prostatectomy prior to start of androgen deprivation therapy and prior to step 1 registration
* Pathologically (histologically) proven diagnosis of adenocarcinoma of the prostate as confirmed at time of prostatectomy; prostatectomy must have been performed within 365 days (1 year) prior to step 1 registrationand any type of radical prostatectomy is permitted, including retropubic, perineal, laparoscopic or robotically assisted; (please note: Prior ablative treatment for benign prostatic hypertrophy or focal high-intensity focused ultrasound therapy [HIFU] prior to prostatectomy is allowed)
* Surgical formalin-fixed paraffin-embedded (FFPE) specimen must be available for submission to GenomeDx for genomic analysis on DECIPHER GRID platform

  * Please note: If a patient already has a Decipher risk score and meets all of the other eligibility criteria, the patient is eligible to be registered; however, the Decipher risk report will need to be submitted to GenomeDx for validation
* Prior androgen deprivation (luteinizing hormone-releasing hormone [LHRH] agonist and/or non-steroidal anti-androgen) is allowed if:

  * Androgen deprivation therapy was initiated within 30 days prior to study enrollment
  * Androgen deprivation therapy was given for ≤ 90 days duration prior to radical prostatectomy
  * Please note: Finasteride or dutasteride must be stopped before treatment but should not determine eligibility
* Pathologically lymph node negative by pelvic lymphadenectomy (pN0) or lymph node status pathologically unknown (undissected pelvic lymph nodes [pNx])
* Any pT-stage based on American Joint Committee on Cancer 7th edition eligible; study entry will be based on the following diagnostic workup:

  * History/physical examination within 60 days prior to step 1 registration
  * Negative distant metastatic workup:

    * A computed tomography (CT) scan of the abdomen and pelvis (with contrast [CT without contrast is permitted if the patient is not a candidate for contrast, i.e., renal function or allergy]) or magnetic resonance imaging (MRI) of the pelvis within 120 days prior to step 1 registration; (Please note: Lymph nodes will be considered negative (NO)if they are =< 1.5 cm short axis);
    * Bone scan within 120 days prior to step 1 registration; (please note: a sodium fluoride [NaF] positron emission tomography [PET]/CT is an acceptable substitute and if the bone scan is suspicious, a plain x-ray, CT scan, NaF PET/CT and/or MRI must be obtained to rule out metastasis; Axumin scans are not allowed for determination of eligibility [e.g. a positive Axumin can in the setting of negative bonescan and CT does not exclude a patient from being eligible for enrollment]).
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1 within 60 days prior to step 1 registration
* Platelets >= 100,000 cell/mm^3 (within 60 days prior to step 1 registration based upon a complete blood count [CBC])
* Hemoglobin >= 10.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 10.0 g/dl is NOT allowed) (within 60 days prior to step 1 registration based upon a CBC)
* Absolute neutrophil count >= 1500 cells/mm^3 (within 60 days prior to step 1 registration based upon a CBC)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 1.5 x the upper limit of normal (within 60 days prior to step 1 registration)
* Total bilirubin (=< 1.5 mg/dl) normal unless history of Gilbert's syndrome (within 60 days prior to step 1 registration)
* The patient or a legally authorized representative must provide study-specific informed consent prior to step 1 registration

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease
* Prior invasive malignancy (except non-melanomatous skin cancer or other in-situ malignancies, or stage Ta bladder cancer) unless disease free for a minimum of 2 years
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable if completed more than two years prior to step 1 registration; prior androgen deprivation is allowed
* Prior whole gland ablative therapy (i.e. cryoablation or high intensity focused ultrasound [HIFU]) for prostate cancer is not allowed
* Prostatectomy performed greater than 365 days (1 year) prior to step 1 registration
* Severe and/or active co-morbidity defined as follows:

  * History of inflammatory bowel disease
  * History of active hepatitis B or C; blood tests are not required to determine if the patient has had hepatitis B or C, unless the patient reports a history of hepatitis
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of step 1 registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization within 15 days of step 1 registration or precluding study therapy at the time of step 1 registration
  * Uncontrolled severe illness or medical condition (including uncontrolled diabetes), which in the judgment of the treating physician would make the administration of chemotherapy inadvisable
* Human immunodeficiency virus (HIV) positive with cluster of differentiation 4 (CD4) count < 200 cells/microliter; note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter within 30 days prior to step 1 registration; note also that HIV testing is not required for eligibility for this protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Freedom from progression (FFP) (Phase II) | From time of randomization to first event, assessed up to 43 months
  Will be determined with a one-sided stratified log-rank test when 89 FFP events have been observed. Both unadjusted and adjusted hazard ratios and the respective 95% confidence interval will be computed. Events for FFP will be the first occurrence of biochemical failure by prostate specific antigen (PSA) >= 0.4 ng/ml over the nadir PSA confirmed by a second PSA higher than the first by any amount, recurrence (local, regional or distant), institution of secondary androgen deprivation therapy and death from any cause.
Metastasis free survival (MFS) (Phase III) | From time of randomization to first occurrence of distant metastasis or death from any cause, assessed up to 9.5 years
  Will be measured with a one-sided stratified log-rank test when 282 MFS events have been observed. Both unadjusted and adjusted hazard ratios and the respective 95% confidence interval will be computed.

SECONDARY OUTCOMES:
Overall survival | Time to death from any cause assessed up to 2.5 years
  Will be analyzed using log-rank methodology and Cox proportional models. Tests for violations of proportionality will performed for the survival models. Fine and Gray's regression also will be used. Both unadjusted and adjusted hazard ratios and the respective 95% confidence interval will be computed.
Time to local progression | Baseline to local or regional recurrence ignoring biochemical failure and distant recurrence and censoring for death, assessed up to 2.5 years
  Both unadjusted and adjusted hazard ratios and the respective 95% confidence interval will be computed.
Proportion of undetectable prostate specific antigen (PSA) with a non-castrate testosterone | At 2.5 years
  Both unadjusted and adjusted hazard ratios and the respective 95% confidence interval will be computed.
Incidence of acute adverse events scored according to the Cancer Therapy Evaluation Program active version of the Common Terminology Criteria for Adverse Events | Up to 30 days post radiation therapy
  Will be compared to late grade 3+ adverse events. Univariate logistic regression will be used to model the distribution of acute adverse events. Multiple logistic regression will be used to model the distribution of acute adverse events adjusted for covariates. Both unadjusted and adjusted odds ratios and the respective 95% confidence interval will be computed and tested using a one-sided Chi-Square test statistic with the significance level of 0.025. Both unadjusted and adjusted hazard ratios and the respective 95% confidence interval will be computed.
Genomic profiling in making adjuvant therapy decisions | Up to 9 years
  Both unadjusted and adjusted hazard ratios and the respective 95% confidence interval will be computed.
Late grade 3+ adverse events scored according to the Cancer Therapy Evaluation Program active version of the Common Terminology Criteria for Adverse Events | From protocol treatment starts to the worst late grade 3+ adverse event, assessed up to 9 years
  Will be compared to acute adverse events. A Fine and Gray's regression model will be used to compare the treatment differences of time to late adverse event with and without adjusting for other covariates. Both unadjusted and adjusted odds ratios and the respective 95% confidence interval will be computed and tested using a one-sided. Will be estimated using the cause-specific hazard rate approach and tested using a significance level of 0.025. Both unadjusted and adjusted hazard ratios and the respective 95% confidence interval will be computed. At least the treatment arm, age, and race (as appropriate) will be considered when it is adjusted in the analysis.

OTHER OUTCOMES:
DECIPHER signature in predicting response | Up to 9 years
  Proposed and additional future translational studies will be assessed following completion of accrual and sample collection. Transcriptomic information generated with the DECIPHER GRID will be used to assess other biologically-relevant question including characterizing the transcriptomic landscape of prostate cancer from younger vs older patients, interrogating the noncoding aspects of the prostate cancer transcriptome, and identifying outcomes based on the molecular subtypes of prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Hurwitz, Principal Investigator — NRG Oncology
Locations (313):
- United States (311):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Adventist Health Cancer Care Center Chico, Chico, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Naval Medical Center -San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - GenesisCare USA - Aventura FP, Aventura, Florida
  - GenesisCare USA - Aventura, Aventura, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - AdventHealth Celebration, Celebration, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - GenesisCare USA - Key West, Key West, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - GenesisCare USA - Lakewood Ranch, Lakewood Rch, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Alton Memorial Hospital, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta, Canada
- Centro Comprensivo de Cancer de UPR, San Juan, Puerto Rico